CLINICAL TRIAL: NCT02081443
Title: In Vitro Pharmacodynamic Effects of Cangrelor on Platelet P2Y12 Receptor Mediated Signaling in Ticagrelor Treated Patients
Brief Title: In Vitro Pharmacodynamic Effects of Cangrelor in Ticagrelor Treated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CIT
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2017-03-03 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; platelet function; ticagrelor; cangrelor
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor 180mg (Experimental): The proposed study will have a prospective, randomized, parallel design in which patients on chronic ticagrelor therapy will be assigned to receive a reloading dose of 90 or 180 mg ticagrelor. Platelet function assays will be done following in vitro incubation with and without 500 nM cangrelor.
  Interventions: Drug: Ticagrelor 90mg
- Ticagrelor 90mg (Active Comparator): The proposed study will have a prospective, randomized, parallel design in which patients on chronic ticagrelor therapy will be assigned to receive a reloading dose of 90 or 180 mg ticagrelor. Platelet function assays will be done following in vitro incubation with and without 500 nM cangrelor.
  Interventions: Drug: Ticagrelor 180mg

INTERVENTIONS:
Drug: Ticagrelor 180mg — The proposed study will have a prospective, randomized, parallel design in which patients on chronic ticagrelor therapy will be assigned to receive a reloading dose of 90 or 180 mg ticagrelor. Platelet function assays will be done following in vitro incubation with and without 500 nM cangrelor.
  Other Names: Brilinta
  Arms: Ticagrelor 90mg
Drug: Ticagrelor 90mg — The proposed study will have a prospective, randomized, parallel design in which patients on chronic ticagrelor therapy will be assigned to receive a reloading dose of 90 or 180 mg ticagrelor. Platelet function assays will be done following in vitro incubation with and without 500 nM cangrelor.
  Other Names: Brilinta
  Arms: Ticagrelor 180mg

SUMMARY:
Cangrelor is a potent intravenous P2Y12 receptor inhibitor with rapid onset and offset of action associated with a greater reduction in ischemic events, including stent thrombosis, in patients undergoing stent procedures who have not been pretreated with clopidogrel. In vitro investigations have shown cangrelor to be associated with more rapid, potent, and consistent platelet inhibition in patients on maintenance prasugrel therapy exposed to a re-loading dose of prasugrel. However, if cangrelor exerts similar effects in ticagrelor treated patients remain unknown. The aim of the present study is to evaluate the effects on platelet function achieved after in vitro incubation with cangrelor in patients on ticagrelor maintenance dose who receive a loading dose of ticagrelor.

DETAILED DESCRIPTION:
A higher degree of platelet inhibition remains the goal in the peri-interventional period in patients undergoing percutaneous coronary interventions (PCI) as this is associated with a lower rate of adverse ischemic events. Ticagrelor and prasugrel are novel and potent generation oral P2Y12 receptor inhibitors associated with a greater reduction in ischemic events compared with clopidogrel. However, both prasugrel and ticagrelor have recently showed variability in pharmacodynamic (PD) response, particularly in patients with ST-elevation myocardial infarction (STEMI) undergoing primary PCI, exposing these patients to an increased risk of thrombotic complications. These findings support the need for intravenous agents with more rapid platelet inhibiting effects. Cangrelor is a potent intravenous P2Y12 receptor inhibitor with rapid onset and offset of action associated with a greater reduction in ischemic events, including stent thrombosis, in patients undergoing PCI who have not been pretreated with clopidogrel. In vitro PD investigations have shown cangrelor to be associated with more rapid, potent, and consistent platelet inhibition in patients on maintenance prasugrel therapy exposed to a re-loading dose of prasugrel. However, if cangrelor exerts similar effects in ticagrelor treated patients remain unknown. The aim of the present study is to evaluate the PD effects achieved after in vitro incubation with cangrelor in patients on ticagrelor maintenance dose who receive a loading dose of ticagrelor. The proposed study will have a prospective, randomized, parallel design in which patients on chronic ticagrelor therapy will be assigned to receive a reloading dose of 90 or 180 mg ticagrelor. PD assessments will be done before and after incubation with cangrelor at 3 time-points. The study hypothesis is that in vitro incubation with cangrelor will lead to incremental P2Y12 receptor blockade, the extent of which will be inversely related to dose of ticagrelor.

ELIGIBILITY:
Inclusion criteria:

1. Patients with angiographically documented coronary artery disease.
2. Age between 18 to 80 years
3. On treatment per standard of care with ticagrelor 90mg/b.i.d. and aspirin <100mg/day for at least 14 days.

Exclusion criteria

1. History of intracranial bleeding
2. Known severe hepatic dysfunction
3. Known hypersensitivy
4. Active bleeding or propensity to bleed
5. Platelet count <80x106/mL
6. Hemodynamic instability
7. Serum creatinine <30 mL/min
8. Use of oral anticoagulants (Vitamin K antagonist, dabigatran, rivaroxaban, apixaban)
9. Recent (<14 days) antiplatelet treatment with a glycoprotein IIb/IIIa inhibitor
10. Blood dyscrasia
11. Patients with sick sinus syndrome (SSS) or II or III degree AV block without pacemaker
12. Drugs interfering CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromicin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir and telithromizycin
13. Hemoglobin < 10g/dL
14. Pregnant females [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study].

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, Principal Investigator — University of Florida
Locations (1):
- Dominick Angiolillo, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from October 2014 to October 2015. Patients were screened and recruited in the Cardiology clinics of the Division of Cardiology of University of Florida Jacksonville.
Pre-assignment Details: 64 patients were consented for the study. Of these, 3 withdrew from the study before being randomized, 1 had an exclusion criteria. A total of 60 patients were randomized to receive study medications.
Groups:
- Ticagrelor 180mg: The proposed study have a prospective, randomized, parallel design in which patients on chronic ticagrelor therapy were randomly assigned to receive a reloading dose of 90 or 180 mg ticagrelor. Platelet function assays was done following in vitro incubation with and without 500 nM cangrelor.
- Ticagrelor 90mg: The proposed study has a prospective, randomized, parallel design in which patients on chronic ticagrelor therapy were randomly assigned to receive a reloading dose of 90 or 180 mg ticagrelor. Platelet function assays were done following in vitro incubation with and without 500 nM cangrelor.
Period: Overall Study
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9) | 57 (8) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 19 | 21 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 21 | 24 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Index (PRI) Determined by Whole Blood Vasodilator-stimulated Phosphoprotein (VASP)
Description: PRI determined by VASP between before and after incubation with 500 nM Cangrelor in each arm of treatment
Time Frame: Baseline
Measure: Mean (Standard Error); unit: %PRI
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Number analyzed (Participants) | 30 | 30
%PRI
  Without cangrelor | 30 (3.6) | 30 (4)
  With cangrelor | 18 (1.7) | 17 (1.8)

2. Secondary Outcome: PRI Measured by VASP
Description: PRI determined by VASP between before and after incubation with 500 nM Cangrelor in each arm of treatment
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: %PRI
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Number analyzed (Participants) | 30 | 30
%PRI
  Without cangrelor | 20 (2.4) | 29 (3.4)
  With cangrelor | 12 (1.6) | 16 (1.5)

3. Secondary Outcome: PRI Measured by VASP
Description: PRI determined by VASP between before and after incubation with 500 nM Cangrelor in each arm of treatment
Time Frame: 4 hours
Measure: Mean (Standard Error); unit: %PRI
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Number analyzed (Participants) | 30 | 30
%PRI
  Without cangrelor | 22 (2.4) | 22 (2)
  With cangrelor | 14 (1.2) | 17 (1.9)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Ticagrelor 180mg | Ticagrelor 90mg
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 180mg (N=30) | Ticagrelor 90mg (N=30)
Dehydration (General disorders) | 1 (1) | 0 (0) — Not study related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes